CLINICAL TRIAL: NCT06924346
Title: Efficacy of Exercise Snacks in Real-World Settings in Individuals Living With Obesity
Brief Title: Exercise Snacks in Obesity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: McMaster University (Other)
Responsible Party: Principal Investigator, Jonathan Little, professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H24-OB-snacks
Record Dates: First submitted 2025-03-26; First posted 2025-04-11 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Snacks (Experimental): Vigorous-intensity bodyweight exercises performed 4 times per day on at least 5 days per week.
  Interventions: Other: Exercise Snacks
- Placebo Exercise (Active Comparator): Low-intensity stretching exercises performed 4 times per day on at least 5 days per week.
  Interventions: Other: Placebo Exercise

INTERVENTIONS:
Other: Exercise Snacks — The "movement breaks" will be individualized to exercise preferences and physical abilities (e.g., fitness, musculoskeletal issues) and adaptable to multiple environments (e.g., home, work) delivered via mobile phone application. Participants will be encouraged to incorporate the movement breaks into their daily schedule based on baseline exercise counselling.
  Arms: Exercise Snacks
Other: Placebo Exercise — The "movement breaks" will be individualized to exercise preferences and physical abilities (e.g., fitness, musculoskeletal issues) and adaptable to multiple environments (e.g., home, work) delivered via mobile phone application. Participants will be encouraged to incorporate the movement breaks into their daily schedule based on baseline exercise counselling.
  Arms: Placebo Exercise

SUMMARY:
To conduct a randomized control trial to determine the feasibility and preliminary efficacy of a 12-week technology-enabled exercise snacks intervention with behaviour change counselling for improving cardiorespiratory fitness and various markers of cardiometabolic health in previously inactive adults living with obesity.

DETAILED DESCRIPTION:
Participants will be randomized into an Exercise Snacks or a Placebo Exercise group for 12 weeks. The former will involve bodyweight exercises performed with vigorous effort and the latter will involve low-intensity stretching and mobility exercises. Following baseline testing, individualized interventions will be delivered via a customized mobile application ("app") or web platform. Participants will be instructed to perform a minimum of 4 isolated bouts of prescribed exercises per day on at least 5 days per week. Each bout will be one minute in duration. The interventions will be individualized and consider exercise preferences and physical abilities (e.g., fitness, musculoskeletal issues), and be adaptable to multiple environments (e.g., home, work). To facilitate this, participants will have a pre-intervention meeting wherein any physical limitations will be documented, and a research assistant trained in health behaviour change techniques will provide a brief exercise counselling session designed to individualize the intervention to the participant's preferences, abilities, and lifestyle. After 12 weeks, participants will be asked to return to the lab for follow-up testing.

ELIGIBILITY:
Inclusion Criteria:

* Aged 35-64 years.
* Habitually engaging in < 150 min moderate-to-vigorous physical activity per week.
* Body mass index 30-45 kg/m2 or 27.5-45 for participants who self-identify as being of Asian or Southeast Asian origin.
* Waist circumference: >88cm for females and >102cm for males, or >80 cm for females and >90 cm for male participants who self-identify as being of Asian or Southeast Asian.
* Not currently diagnosed with a cardiometabolic disease (e.g., coronary artery disease, stroke, diabetes, non-alcoholic fatty liver disease).
* Taking ≤2 commonly prescribed medications for the prevention of cardiometabolic diseases (e.g., statins, antihypertensives).
* Not a current smoker
* Cleared to engage in physical activity using the Get Active Questionnaire and, if applicable, consultation with a health care provider or Qualified Exercise Professional.
* Access to a computer, tablet or smartphone for intervention delivery and tracking.
* Ability to read and write in English.

Exclusion Criteria:

* Chronic musculoskeletal condition or recent (within 2 years) cardiovascular event preventing participation in exercise.
* Lack of internet access.
* Angina upon exertion assessed by the Rose Angina Questionnaire.
* Prescribed beta-blockers that can compromise the validity of heart rate measurements. during the exercise test.
* Have a scheduled surgical procedure within the next 3-4 months that would prevent exercise participation.
* Currently participating in another clinical trial that interferes with the study procedures.
* Currently pregnant or planning on becoming pregnant during the intervention (i.e., within the next 4 months).
* Uncontrolled high blood pressure (>160/90 mmHg)

Ages: 35 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-07-14 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Determine the number of individuals living with obesity that are eligible to participate in the trial | through study completion, an average of 18 months
  The number of participants approached and reasons for not joining the study.
Determine the number of eligible participants who would be willing to take part in this trial | through study completion, an average of 18 months
  The number of participants who enroll.
Determine the number and percentage of participants retained after the 12-week intervention | after the 12-week intervention
  Number and percentage of participants who drop-out and reasons.
Determine the number of one-minute exercise bouts performed during the 12-week intervention | during the 12 weeks
  Number of exercise bouts performed each week of the intervention.

SECONDARY OUTCOMES:
Change in cardiorespiratory fitness measured before and after the 12-week intervention | 0-12 weeks
  Cardiorespiratory fitness will be measured using an incremental exercise test on a motorized treadmill at baseline and after the 12-week intervention.
Change in lower body muscular endurance before and after the 12-week intervention | 0-12 weeks
  The 30-second sit-to-stand will be measured at baseline and after the 12-week intervention.
Change in upper body maximal strength before and after the 12-week intervention | 0-12 weeks
  Grip strength test using a hand dynamometer will be measured at baseline and after the 12-week intervention.
Change in waist circumference before and after the 12-week intervention | 0-12 weeks
  Waist circumference will be measured at baseline and after the 12-week intervention.
Change in weight before and after the 12-week intervention | 0-12 weeks
  Weight will be measured at baseline and after the 12-week intervention.
Change in body mass index before and after the 12-week intervention | 0-12 weeks
  Body mass index will be measured at baseline and after the 12-week intervention.
Change in fasting glucose measured before and after the 12-week intervention | 0-12 weeks
  Fasting glucose will be measured at baseline and after the 12-week intervention.
Change in fasting insulin measured before and after the 12-week intervention | 0-12 weeks
  Fasting insulin will be measured at baseline and after the 12-week intervention.
Change in systolic blood pressure measured before and after the 12-week intervention | 0-12 weeks
  Seated systolic blood pressure will be measured at baseline and after the 12-week intervention.
Change in diastolic blood pressure measured before and after the 12-week intervention | 0-12 weeks
  Seated diastolic blood pressure will be measured at baseline and after the 12-week intervention.
Change in physical activity assessed during the first and last weeks of the intervention | weeks 0 and 12
  Physical activity measured using accelerometry during week 0 and week 12.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - University of British Columbia Okanagan, Kelowna, British Columbia
  - McMaster University, Hamilton, Ontario

IPD SHARING:
Plan to Share IPD: No